CLINICAL TRIAL: NCT02510157
Title: Effect of Dexamethasone on the Action of Sugammadex
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Attikon Hospital (Other)
Responsible Party: Principal Investigator, Chrysanthi Batistaki, Assistant Professor of Anesthesiology, 2nd Department of Anesthesiology, School of Medicine, University of Athens, Greece, Attikon Hospital
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 711/19-3-15
Record Dates: First submitted 2015-05-16; First posted 2015-07-29 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-07

CONDITIONS: Neuromuscular Blockade
Keywords: sugammadex; dexamethasone; neuromuscular blockade
MeSH Terms: interventions — Dexamethasone; Saline Solution; Sugammadex

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- dexamethasone (Active Comparator): Dexamethasone is administered intravenously before induction of anaesthesia. Deep neuromuscular blockade is induced with rocuronium and is assessed by acceleromyography (post-tetanic count stimulation) on the ulnar nerve of the patient's hand. At the end of surgery, sugammadex 4 mg/kg is administered to reverse neuromuscular blockade.
  Interventions: Drug: Dexamethasone; Drug: sugammadex
- normal saline (Placebo Comparator): Normal saline is administered intravenously before induction of anaesthesia. Deep neuromuscular blockade is induced with rocuronium and is assessed by acceleromyography (post-tetanic count stimulation) on the ulnar nerve of the patient's hand. At the end of surgery, sugammadex 4 mg/kg is administered to reverse neuromuscular blockade.
  Interventions: Drug: Normal Saline; Drug: sugammadex

INTERVENTIONS:
Drug: Dexamethasone — active comparator
  Arms: dexamethasone
Drug: Normal Saline — placebo controlled intervention
  Other Names: N/S 0.9%
  Arms: normal saline
Drug: sugammadex — sugammadex is administered in both groups to reverse deep neuromuscular blockade at the end of surgery

SUMMARY:
This study aims to investigate the possible clinical effect of dexamethasone on the action of sugammadex when it is administered to reverse deep neuromuscular blockade caused by rocuronium in laparoscopic cholecystectomies.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-70 years
* laparoscopic cholecystectomy
* operation < 3 hours

Exclusion Criteria:

* age <18 or >70 years old
* ASA physical status >3
* central nervous system diseases
* severe psychiatric disorders under treatment
* cognitive dysfunction
* known or suspected allergy to the administered drugs
* operations > 3 hours
* surgical intraoperative complications-open cholecystectomy
* severe renal or liver disease
* diabetes melitus
* immunosuppressed patients
* chronic immunosuppresant therapy (corticosteroids or other drugs)
* all contraindications to corticosteroids administration
* patiens on chronic use of opioids

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Time to train-of-four (TOF) ratio of 0.9 since administration of sugammadex | minutes after administration of sugammadex (0 to 30 minutes)
  measurement of time after administration of the reversal agent (sugammadex) to achieve train-of-four (TOF0 ratio of 0.9 (up to 30 minutes)

SECONDARY OUTCOMES:
Postoperative pain | 1, 6, 12, 24 hours postoperatively
  Assessed by Numeric Rating Scale 0-10
Postoperative nausea and vomiting | 1, 6, 12, 24 hours postoperatively
  Assessed by nausea/vomiting scale (11. Myles PS, Wengritzky R. Simplified postoperative nausea and vomiting impact scale for audit and post-discharge review. Br J Anaesth 2012; 108: 423-429)

OTHER OUTCOMES:
Time from end of surgery to extubation of patient | minutes after administration of sugammadex (0 to 30 minutes)
  measurement of time after administration of the reversal agent (sugammadex) to achieve extubation of patient (up to 30 minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Department of Anesthesiology, Attikon Hospital, 1 Rimini str., Athens, Greece